CLINICAL TRIAL: NCT02238691
Title: Risk of Gastric Insufflation Related to Facemask Ventilation Technique During Anaesthetic Induction
Brief Title: Risk of Gastric Insufflation Related to Facemask Ventilation Technique During Anaesthetic Induction, With or Without PEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Alex de Leon, PhD, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pelles PEEP-studie
Record Dates: First submitted 2014-08-13; First posted 2014-09-12 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Air Insufflation; Regurgitation
Keywords: PEEP; Air insufflation; Mask ventilation; Esophageal manometry; Esophageal impedance
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mask ventilation with PEEP (Experimental): 15 subjects will undergo anesthetic induction with application of PEEP of 10 cm H2O during mask ventilation.
  Interventions: Procedure: Mask ventilation with PEEP via a face mask device
- Mask ventilation without PEEP (No Intervention): 15 subjects will undergo anesthetic induction without PEEP during mask ventilation.

INTERVENTIONS:
Procedure: Mask ventilation with PEEP via a face mask device — 15 subjects will undergo anesthetic induction with an application of PEEP of 10 cm H2O during mask ventilation via a face mask.
  15 subjects will undergo anesthetic induction without PEEP during mask ventilation via a face mask.
  Arms: Mask ventilation with PEEP

SUMMARY:
Continuous positive pressure during anesthetic induction is today not routinely used partly a to the risk of gastric insufflation because of higher ventilatory pressures. However there are conflicting data with improvement of GERD symptoms in CPAP treated OSA patients. The investigators aim to compare the risk of gastric insufflation regarding mask ventilation technique, with or without positive end expiratory pressure. For measurements a High Resolution Impedance Manometry Catheter is used.

DETAILED DESCRIPTION:
Anesthetic induction agents cause a number of physiological changes within the respiratory system. Almost every induction agent causes apnoea. There is a reduction of FRC and an increase in airway resistance. Combined with preoxygenation with a high fraction of oxygen there is a significant risk of pulmonary atelectasis. Adding a continuous positive pressure during ventilation of the apnoeic patient improves many of the respiratory effects caused by induction agents. However the added continuous pressure will increase the total inspiratory pressure and a high inspiratory pressure is associated with an increased risk of gastric insufflation during mask ventilation. On the other hand there are data suggesting that continuous positive pressure is beneficial in treatment of GERD-symptoms.

The investigators hypothesis is, if performed correctly, that the continuous positive pressure will not increase the risk of gastric insufflation. In order to investigate this matter 30 healthy human subjects will undergo anesthetic induction, 15 with no PEEP added and 15 with a PEEP of 10 cm H2O during mask ventilation.

Protocol:

1. Preoxygenation, 100 % oxygen via Face mask for 3 minutes with 0 PEEP or 10 cm H2O PEEP.
2. Start of Remifentanil Target Controlled Infusion, target concentration 6 ng/ml.
3. Propofol 2-2.5mg/kg to adequate depth of anesthesia.
4. 30 seconds after apnea mask ventilation with Dräger ZEUS IE starting with an inspiratory pressure of 3cm H2O that is gradually increased to a maximum of 30 cm H20 or to signs of air insufflation in the esophagus. Group 1 with 0 PEEP and group 2 with 10 cm H2O PEEP.
5. End of Remifentanil- and Propofol infusion.

Pressures and passage of air or liquid from pharynx to stomach will be continuously registered during the procedure. For measurements a High Resolution Impedance Manometry Catheter with the ability to measure pressures and impedance simultaneously will be used.

The esophagus and the stomach is divided into four functional units for analysis.

1. The upper esophageal sphincter
2. The esophageal body (3 cm below upper esophageal sphincter to 3 cm over the lower esophageal sphincter)
3. The lower esophageal sphincter
4. The stomach (3 cm below the lower esophageal sphincter)

The different units are detected in pressure plots where the levels of pressure reflects the anatomical units. Manometric values is specified in mmHg. For detection of passage of air and flow of liquid an impedance baseline is set before measurements start. Passage of air is defined as a sudden rise in impedance of 1 kΩ in anterograde direction. Detection of fluid is defined as a 50% decline in impedance. For analysis of data Mano View analysis software is used.

Pressures and impedance will be continuously recorded during the time frame from preoxygenation to maximum inspiratory pressures are reached. Data will be analysed at each level of pressure 3, 5, 10, 15, 20, 25 and 30 cm H2O. Contained data will be statistically compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18-40 years
* Signed and informed consent
* Subject will and is assumed to be able to follow protocol

Exclusion Criteria:

* Known gastro intestinal/heart/lung/kidney or neurological disease
* Use of drugs that interfere with esophageal motility
* Diabetes
* Pregnancy or breastfeeding
* BMI >30

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Level of inspiratory pressure for gastric insufflation | One hour

SECONDARY OUTCOMES:
Pressure changes in the esophagus related to ventilation technique. | One hour

OTHER OUTCOMES:
Pressure changes in the stomach after gastric insufflation | One hour

CONTACTS AND LOCATIONS:
Overall Officials: Alex deLeon, MD, Phd, Principal Investigator — Region Örebro County
Locations (1):
- Örebro University Hospital, Örebro, Sweden

REFERENCES:
- [Derived] Cajander P, Edmark L, Ahlstrand R, Magnuson A, de Leon A. Effect of positive end-expiratory pressure on gastric insufflation during induction of anaesthesia when using pressure-controlled ventilation via a face mask: A randomised controlled trial. Eur J Anaesthesiol. 2019 Sep;36(9):625-632. doi: 10.1097/EJA.0000000000001016. PMID 31116114